CLINICAL TRIAL: NCT00387634
Title: A Phase IV, Uncontrolled, Open-label, Single-center Study in Adolescents and Adults: Evaluation of Immunogenicity and Safety of the First Booster Immunization With Novartis' TBE Vaccine for Adults in Participants of Study V48P7 and Long-term Evaluation of Immunogenicity up to 5 Years After First Booster Immunization
Brief Title: Safety and Long-term Evaluation (up to 5 Years) of First Booster Immunization With Novartis' TBE Vaccine for Adults in Adolescents and Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V48P7E1
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Tick Born Encephalitis
Keywords: tick born encephalitis, TBE, adults

ARMS (4):
- Arm 1 (Active Comparator): Blood draw only, no vaccine
  Interventions: Biological: TBE vaccine for adults
- Arm 2 (Active Comparator): Blood draw only, no vaccine
  Interventions: Biological: TBE vaccine for adults
- Arm 3 (Active Comparator): Blood draw only, no vaccine
  Interventions: Biological: TBE vaccine for adults
- Arm 4 (Active Comparator): Blood draw only, no vaccine
  Interventions: Biological: TBE vaccine for adults

INTERVENTIONS:
Biological: TBE vaccine for adults — Serology blood draw.

SUMMARY:
evaluate safety and immunogenicity of first TBE booster and long-term immunogenicity up to 5 years after first TBE booster

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects who have completed study V48P7

Exclusion Criteria:

* acute illness at day of immunization
* general decrease in resistance
* progressive neurological disorders
* history of febrile or afebrile convulsions
* major congenital defects
* serious chronic illness
* hypersensitivity to study vaccine
* treatment with immunosuppressants or systemic corticosteroids, immunoglobulins, whole blood or plasma derivates

Ages: 15 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2006-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
immunogenicity of TBE vaccine for adults when given as first booster dose as measured by neutralisation test and ELISA | On day 21, year 1, year 2, year 3, year 4, year 5

SECONDARY OUTCOMES:
safety of TBE vaccine for adults with respect to local and systemic reactions and adverse event reporting | Local and systemic reactions: up to Day 3 post vaccination; Adverse events: 21 days post vaccination; SAEs: throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Study Chair — Novartis
Locations (1):
- Hradec Králové, Czechia

REFERENCES:
- [Derived] Beran J, Xie F, Zent O. Five year follow-up after a first booster vaccination against tick-borne encephalitis following different primary vaccination schedules demonstrates long-term antibody persistence and safety. Vaccine. 2014 Jul 23;32(34):4275-80. doi: 10.1016/j.vaccine.2014.06.028. Epub 2014 Jun 17. PMID 24950352